CLINICAL TRIAL: NCT02374424
Title: Phase II Study With Ga101-DHAP as Induction Therapy in Relapsed/Refractory Diffuse Large B-cell Lymphoma (DLBCL) Patients Before High-Dose Chemotherapy BEAM With Autologous Stem Cell Transplantation (ASCT)
Brief Title: Phase II Study With Ga101-DHAP as Induction Therapy in Relapsed/Refractory DLBCL Patients
Acronym: GIOTTO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis planned as per protocol didn't provide positive outcome therefore enrollment was not reopened. However, the enrolled patients concluded therapy and continued into the follow-up phase. The study was closed only after LVLP.
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_GA101_DHAP
Record Dates: First submitted 2015-02-17; First posted 2015-02-27 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Diffuse, Large B-Cell, Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GA101_DHAP (Experimental): Patients receive: GA101-DHAP x 2, restaging, mobilization and collection of peripheral blood stem cells, + GA101-DHAP x 2, restaging with PET and CT and consolidation with BEAM and ASCT in patients in response (CR+PR).
  During the treatment period of four cycles, all patients will receive a total of four 28-day courses of chemotherapy.
  Interventions: Drug: GA101_DHAP

INTERVENTIONS:
Drug: GA101_DHAP — Aim of the study is to assess whether the addition of GA101 to DHAP is more promising than standard R-DHAP, as induction therapy before high dose chemotherapy BEAM with ASCT with respect to response.
  Scheme of treatment:
  * GA101 1000 mg iv day 1, 8, 15 on first cycle (starting from cycle 2, GA101 1000 mg day 1)
  * Cisplatin 100 mg/sqm iv day 1 of every cycles in 24-hours infusion
  * Cytarabine 2000 mg/sqm in 3-hours infusion every 12 hours iv day 2 of every cycles
  * Dexamethasone 40 mg day 1-4 of every cycles
  * Pegfilgrastim 6 mg sc single dose 24 hours after the end of chemotherapy or G-CSF from day 4 till stem cell harvest during mobilization's course (II o III cycle GA101-DHAP)
  * GA101 1000 mg iv 24 hours before apheresis as purging in vivo during second courses of therapy

SUMMARY:
Aim of this trial is to assess the efficacy of new anti-CD20 antibody (GA101) in association with DHAP as induction therapy before high dose chemotherapy BEAM with ASCT in patients with relapsed/refractory DLBCL.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single arm, phase II trial in young patients (18-65 years) affected by relapsed/refractory Diffuse Large B-cell Lymphoma (DLBCL) at diagnosis,eligible to high-dose therapy.

Aim of the study is to assess whether the addition of GA101 to DHAP is more promising than standard R-DHAP, as induction therapy before high dose chemotherapy BEAM with ASCT with respect to response.

The study is designed primarily to evaluate the efficacy of GA101-DHAP in patients with DLBCL who have relapsed or are refractory to one chemotherapy regimen and secondarily to assess safety and capability to mobilize peripheral stem cells The study is designed with two stages and with stopping rules after the first stage. In particular, at the end of the first stage, the study will be stopped if the efficacy is too low or if the toxicity, measured during the drug administration period, is too high with respect to pre-defined thresholds. .

ELIGIBILITY:
Inclusion Criteria:

1. 18≥ Age < 65
2. Relapsed/refractory disease after receiving one line of standard R-CHOP like chemotherapy
3. Diffuse Large B-cell Lymphoma at relapse. The re-biopsy is particularly recommended if relapse is over 1 year from previous complete remission. If this is harmful for the patient, the patient can be enrolled if archival tumor sample and block from first diagnosis are available.
4. Measurable and/or evaluable disease
5. Any Ann Arbor stage and IPI group at relapse
6. Performance status < 2 according to Eastern Cooperative Oncology Group (ECOG) scale unless due to lymphoma
7. No Central Nervous System (CNS) disease (meningeal and/or brain involvement by lymphoma)
8. Adequate haematological counts: Absolute Neutrophil Count (ANC) > 1.5 x 109/L, Hgb > 10.5 g/dl (transfusion independent), Platelet count > 75 x 109/L (transfusion independent), with the exception of cytopenia due to lymphoma bone marrow involvement
9. Normal liver function (ALP, AST, ALT, GGT, conjugated bilirubin total < 2 x ULN) if not related to lymphoma
10. Normal kidney function (creatinine clearance >= 80 ml/min)
11. Cardiac ejection fraction > 50% (MUGA scan or echocardiography)
12. Normal lung function
13. Absence of active infections
14. Non peripheral neuropathy or active neurological non neoplastic disease of CNS
15. Non major surgical intervention prior 3 months to randomization if not due to lymphoma and/or not other disease life-threatening that can compromise chemotherapy treatment
16. Disease free of prior malignancies other than lymphoma for > 3 years with exception of currently treated squamous cell and basal cell carcinoma of the skin or carcinoma in situ of the cervix or breast
17. Life expectancy > 6 months
18. No psychiatric illness that precludes understanding concepts of the trial or signing ten informed consent
19. Written informed consent
20. Women must be:

    1. postmenopausal for at least 1 year (must not have had a natural menses for at least 12 months)
    2. surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy),
    3. abstinent (at the discretion of the investigator/per local regulations), or
    4. if sexually active, be practicing a highly effective method of birth control (eg, prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method (eg, condoms, diaphragm, or cervical cap, with spermicidal foam, cream, or gel, male partner sterilization) as local regulations permit, before entry, and must agree to continue to use the same method of contraception throughout the study. They must also be prepared to continue birth control measures for at least 18 months after terminating treatment.
21. Women of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening
22. Men must agree to use an acceptable method of contraception (for themselves or female partners as listed above) for the duration of the study. Men must agree to use a double barrier method of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study drug.

Exclusion Criteria:

1. Diagnosis of Lymphoblastic Lymphoma, Burkitt Lymphoma, Non Hodgkin Lymphoma CD20 negative, Mantle Cell Lymphoma, Follicular Lymphoma, Primary Mediastinal Lymphoma
2. Age ≥ 65 years
3. Patients ineligible to high-dose chemotherapy
4. Performance status > 2 according to ECOG scale if not due to lymphoma
5. Patients who previously received GA101 (obinutuzumab) are excluded.
6. Patient has known or suspected hypersensitivity or intolerance to Rituximab
7. Patient has received an experimental drug or used an experimental medical device within 4 weeks before the planned start of treatment. Concurrent participation in nontreatment studies is allowed, if it will not interfere with participation in this study.
8. CNS disease (meningeal and/or brain involvement by lymphoma)
9. History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances
10. Positive test results for chronic hepatitis B infection (defined as positive HBsAg serology). Patients with occult or prior hepatitis B infection (defined as positive total hepatitis B core antibody and negative HBsAg) may be included if HBV DNA is undetectable. These patients must be willing to undergo monthly DNA testing.
11. Positive test results for hepatitis C (HCV antibody serology testing). Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
12. Known history of HIV seropositive status. For patients with unknown HIV status, HIV testing will be performed at screening if required by local regulations.
13. Uncontrolled diabetes (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months before first dose of study drug
14. Uncontrolled or severe cardiovascular disease including myocardial infarction within six months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis
15. Cardiac ejection fraction < 45% (MUGA scan or echocardiography)
16. Creatinine clearance < 45 ml/min
17. Presence of major neurological disorders
18. Active infection
19. Major surgical intervention prior 3 months to randomization if not due to lymphoma and/or other disease life-threatening that can compromise chemotherapy treatment
20. Prior malignancies other than lymphoma in the last 3 years with exception of currently treated squamous cell and basal cell carcinoma of the skin or carcinoma in situ of the cervix or breast
21. Life expectancy < 6 months
22. Any other coexisting medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent.
23. If female, the patient is pregnant or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Aim of this trial is to assess the efficacy of new anti-CD20 antibody (GA101) in association with DHAP as induction therapy before high dose chemotherapy BEAM with ASCT in patients with relapsed/refractory DLBCL. | 4 months
  Primary objective is to assess whether the treatment achieves an absolute increase of the CR proportion of at least 20% (from 30% to 50%) with respect to the standard treatment.
  The complete response rate (CR) evaluated by PET scan after four cycles of GA101-DHAP before ASCT according to Cheson criteria.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) prior to consolidation with BEAM and ASCT | 2 years
  A patient is defined as a responder if she/he has a complete or partial response, evaluated by PET/TC, after four cycles of GA101-DHAP
Progression free survival (PFS) at 6 month after the end of treatment (EOT) | 6 month
  Measured from the date of starting salvage therapy to the date of disease progression, relapse or death from any cause. Responding patients and patients who are lost to follow up will be surveyed at their last assessment date.
Overall Survival (OS) at 2 years after the EOT | 2 years
  Measured from the date of starting salvage therapy to the date of death from any cause. Patients alive at the time of the final analysis will be surveyed at the date of the last contact. For both PFS and OS minimum follow up time required for all patients will be 2 years.
Toxicity: Severe, life-threatening, fatal (grade 3, 4 and 5) and/or serious adverse events | 2 years
  Severe, life-threatening, fatal (grade 3, 4 and 5) and/or serious adverse events are defined according to "Common Terminology Criteria for Adverse Events" (CTCAE), version 4.0. and adverse events of special interests (AESI)
The hematopoietic cell mobilization | 2 years
  Mobilizing potential: amount of CD34 + stem cell collected /Kg
Feasibility: the rate of patients actually proceeding to ASCT | 2 years
  Proportion of patients successfully completing ASCT

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Martelli, MD, Principal Investigator — Dipartimento di Biotecnologie Cellulari ed Ematologia, "La Sapienza" Roma
Locations (10):
- Italy (10):
  - Ospedale San Bortolo, Vicenza, VI
  - Ospedale di Bolzano, Reparto di Ematologia & CTMO, Bolzano
  - A.O. Universitaria Careggi, Florence
  - Ospedale dell'Angelo, U.O. Ematologia, Mestre
  - A.O. Universitaria Policlinico Di Modena, Modena
  - Ematologia Policlinico San Matteo, Pavia
  - AO di Perugia S. Maria della misericordia, Perugia
  - Ematologia Ospedale S.Camillo Forlanini, Roma
  - Policlinico Umberto I - Università "La Sapienza", Roma
  - Ematologia e Trapianto Istituto Regina Elena IFO, Roma

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT02374424/Prot_SAP_000.pdf